CLINICAL TRIAL: NCT02459366
Title: Study of School and Graduate Institute of Physical Therapy College of Medicine in Taiwan
Brief Title: Correlation of Thoracolumbar Fascia Mechanical Properties and Compensate Mechanisms of Asymmetric Skeletal Muscle
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201412156RINA
Record Dates: First submitted 2015-05-26; First posted 2015-06-02 (Estimated); Last update posted 2015-12-30 (Estimated); Status verified 2015-12

CONDITIONS: Low Back Pain
Keywords: Thoracolumbar fascia; Mechanical properties; Low back pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- control: establish the reliability of measurement of lumbopelvic asymmetry, mechanical and physical properties of thoracolumbar fascia, and the norm of different age
- low back pain: compare the differences among asymptomatic subjects and patients with and without lumbopelvic asymmetry, and investigate whether lumbopelvic symmetry, core muscle contractility, proprioception and standing balance change after manipulating thoracolumbar fascia tissue by physical therapy

SUMMARY:
The objective of three-year research is to investigate the relationship between thoracolumbar fascia tissue characteristics, lumbopelvic asymmetry, core muscle contractility, proprioception and standing balance in different ages of asymptomatic participants and patients with CMLBP.

DETAILED DESCRIPTION:
Background: Chronic myofascial low back pain (CMLBP) is a common musculoskeletal disease. Deep fascia is the structures which insufficient in the theory of spinal stability, the major biomechanical role of the thoracolumbar fascia are segmental control and stability of the spine and sacroiliac joint, its biomechanical role is influenced by its mechanical properties of the fascia. Fascia provide the function of sensation and coordination, it is helpful for discussion the compensatory mechanisms for patients with chronic low back pain, and contribution to the development of appropriate therapeutic strategies or combined treatments in innovative applications. However due to the lack of understanding of myofascia, there are difficulties in diagnosis and treatments. It is necessary to establish methods of assessing fascia and complete series of study for understanding fascia and its attaching muscles.

Objective: The objective of three-year research is to investigate the relationship between thoracolumbar fascia tissue characteristics, lumbopelvic asymmetry, core muscle contractility, proprioception and standing balance in different ages of asymptomatic participants and patients with CMLBP.

Method: 270 subjects are recruited in this study, with ages ranging from 20 to 74 years old. 120 of the subjects are patients with CMLBP and 150 are asymptomatic participants. Instrument in use including real time ultrasound imaging, Zebris 3D motionanalysis system and force plate system. The first year is to establish the reliability of measurement of lumbopelvic asymmetry, mechanical and physical properties of thoracolumbar fascia, and the norm of different age. The second year is to compare the differences among asymptomatic subjects and patients with and without lumbopelvic asymmetry, and investigate whether lumbopelvic symmetry, core muscle contractility, proprioception and standing balance change after manipulating thoracolumbar fascia tissue by physical therapy. The third year is to investigate the treatment effect on chronic myofascial back pain patient after 8 weeks exercise training with the aid of physical agent.

ELIGIBILITY:
Inclusion criteria:

* Asymptomatic subjects
* Age between 20-74 years old
* In the past three months did not feel uncomfortable more than one day on waist region, and did not relapsed more than once within three months

Subjects with chronic low back pain

* Age between 20-74 years old
* In the past three months felt uncomfortable more than one day on waist region, and relapsed more than once within three months
* Visual pain scores (VAS ≧ 3)

Exclusion criteria:

1. Can not communicate clearly with people
2. Any open wounds
3. Any history of cancer or malignancy
4. The bleeding disorders
5. Pregnancy

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: community sample
Sampling Method: Non-Probability Sample
Enrollment: 270 (Estimated)
Dates: Start 2015-05; Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Tissue characteristics of thoracolumbar | 30 minutes

SECONDARY OUTCOMES:
Contraction ability of core muscles | 30 minutes
  using ultrasound image to measure the thickness change of core muscles
The re-position range of motion of lumbar spine | 30 minutes
Scale of standing balance | 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Shwu-Fen Wang, Principal Investigator — NTUH
Locations (1):
- National Taiwan University Hospital, Taipei, Test2, Taiwan